CLINICAL TRIAL: NCT07322315
Title: Diagnostic Value of Transcranial Doppler Ultrasound for Evaluating Neonatal Craniocerebral Injuries
Status: Recruiting | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Neamat Mohamed Kamal Omar, Resident of Diagnostic and Intervention Radiology, Faculty of Medicine, Kafr- Elsheikh University, Kafrelsheikh University
Other Study IDs: KFSIRB200-842
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Diagnostic Value; Transcranial Doppler Ultrasound; Neonatal Craniocerebral Injuries
MeSH Terms: interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: High-risk neonates with confirmed risk factor.
  Interventions: Device: Transcranial Doppler ultrasound
- Group B: Healthy neonates without any identified risk factor, matched to Group A for age and sex.
  Interventions: Device: Transcranial Doppler ultrasound

INTERVENTIONS:
Device: Transcranial Doppler ultrasound — Trans-cranial ultrasound will be carried out for assessment of blood flow velocity in the anterior [ACA] and middle cerebral arteries [MCA] using duplex pulsed Doppler ultrasound.

SUMMARY:
This study aims to evaluate the diagnostic value of transcranial Doppler ultrasonography (TCD) for evaluating neonatal craniocerebral injuries.

DETAILED DESCRIPTION:
A high-risk neonate refers to an infant, irrespective of gestational age or birth weight, who exhibits an elevated likelihood of experiencing health complications or death. Preterm infants, defined as those born alive at a gestational age of less than 37 weeks, have seen increased birth and survival rates due to advancements in medical technology and the widespread establishment of Neonatal Intensive Care Units (NICUs).

Neonatal sepsis is one of the leading causes of morbidity and mortality among term and preterm infants worldwide.

Transcranial Doppler ultrasonography (TCD) is the only noninvasive method that enables reliable evaluation of blood flow in the basal intracerebral vessels, providing physiological information complementary to anatomic imaging. TCD is relatively inexpensive, can be performed at the bedside, and enables monitoring in acute emergency settings and for prolonged periods with high temporal resolution, making it ideal for studying dynamic cerebrovascular responses.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes.
* High-risk neonates with any of the following:

  * Critically ill neonates.
  * Neonatal sepsis.
  * Neonatal encephalopathy includes hypoxic-ischemic encephalopathy.
  * Respiratory distress.
  * Neonatal seizures.
  * Birth asphyxia.
  * Signs and or symptoms of central nervous system disorders like microcephaly, macrocephaly, hypotonia, unexplained poor feeding,
  * Neonates born out of traumatic/instrumental labor.
  * Suspected metabolic disturbances.
  * Neonates with low APGAR score (<7).
  * Neonates with low birth weight (<2.5 kg).

Exclusion Criteria:

* Congenital malformations.
* Genetic metabolic diseases or other severe complications.
* Severe intrauterine infection.

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This prospective observational study will be carried out on 60 neonates admitted to Kafr- Elsheikh University Hospitals over a period of one year starting from approval of the Ethics Committee of Kafr- Elsheikh, Faculty of Medicine and parents of all the included patients will provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of transcranial Doppler ultrasound | 6 months post-procedure
  The sensitivity of transcranial Doppler ultrasound in diagnosing brain injury will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.